CLINICAL TRIAL: NCT06208436
Title: The Survival Outcome of Adjuvant Chemotherapy for Stage I Pancreatic Cancer Stratified by Pathologic Risk Factors
Brief Title: The Survival Outcome of Adjuvant Chemotherapy for Stage I Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Jihui Hao, Professor, Tianjin Medical University Cancer Institute and Hospital
Other Study IDs: Adchmopan01
Record Dates: First submitted 2023-12-25; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Pancreas Cancer; Chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TMUCIH-PDAC: Between 2010 and 2021, the data of patients who underwent surgical resection and were pathologically diagnosed as PDAC from Tianjin Medical University Cancer Institute and Hospital (TMUCIH) were collected retrospectively.
  Interventions: Other: Adjuvant chemotherapy

INTERVENTIONS:
Other: Adjuvant chemotherapy — Patients received adjuvant chemotherapy (5-FU-based or gemcitabine-based regimens) or underwent surgery alone

SUMMARY:
This study aimed to evaluate the impact of adjuvant chemotherapy on survival in patients with Stage I pancreatic cancer stratified by pathologic risk factors.

ELIGIBILITY:
Inclusion Criteria: Patients who underwent surgical resection and were pathologically diagnosed as PDAC between 2010 and 2021.

-

Exclusion Criteria: Patients with pN1-N2, patients with pT3-T4, patients with distant metastasis, patients who received neoadjuvant therapy, patients with R1 resection, and patients who died due to perioperative mortality within 30 days.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage I PDAC patients who underwent radical surgery.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-07 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | January 2010 to February 2023
  The period between surgical resection to the date of recurrence.

SECONDARY OUTCOMES:
Overall survival | January 2010 to February 2023
  The period between surgical resection to the date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Jihui, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No